CLINICAL TRIAL: NCT01109849
Title: Novel Approach to Stimulant Induced Weight Suppression and Its Impact on Growth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH083692 (NIH)
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-06

CONDITIONS: ADHD; Growth
Keywords: ADHD; growth; BMI; stimulant medication
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Behavior Therapy; Methylphenidate; Nurse Clinicians; Central Nervous System Stimulants; Treatment Interruption

STUDY DESIGN:
Intervention Model Description: initial randomization to behavior or extended release stimulant (ER stimulant) arms.
  Participants in either arm meting criteria for a weight recovery intervention (based on change in zBMI) will be adaptively randomized to one of three weight recovery arms (Monitoring, Drug Holiday, Caloric Supplementation)
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- weight recovery treatment- monitoring (Active Comparator): Subjects in either the behavior therapy arm or the medication arm will be assigned to one of 3 treatments if subject does not meet projected BMI goals. In the monitoring arm , participants will continue on their ER stimulant 7 days a week and have their weight, height and BMI checked monthly.
  Interventions: Other: monitoring
- behavior therapy (Active Comparator): 10 week basic parent training, advanced 8 week parent training course. monthly boosters, option for individual parent training sessions, school consultant assigned to each subject
  Interventions: Behavioral: behavior therapy
- ER stimulant (Experimental): daily use of 12 hour extended release methylphenidate product
  Interventions: Drug: Extended release (ER) methylphenidate product
- weight recovery treatment- caloric supplement (Experimental): Subjects in either the behavior therapy arm or the medication arm will be assigned to one of 3 treatments if subject does not meet projected BMI goals. In the caloric supplement arm, participants will continue on their ER stimulant 7 days a week, have their weight, height and BMI checked monthly and be prescribed a 150 kcal caloric supplement to be consumed every evening.
  Interventions: Dietary Supplement: caloric supplement
- weight recovery treatment- drug holiday (Experimental): Subjects in either the behavior therapy arm or the medication arm will be assigned to one of 3 treatments if subject does not meet projected BMI goals. In the drug holiday arm, participants will only take their ER stimulant on school days a week and have their weight, height and BMI checked monthly.
  Interventions: Other: drug holiday

INTERVENTIONS:
Behavioral: behavior therapy — combination of individual and group parent training plus school consultation
  Other Names: behavior modification
  Arms: behavior therapy
Drug: Extended release (ER) methylphenidate product — medication to be taken daily for duration of study unless assigned to weight promotion arm
  Other Names: Concerta, OROS-MPH; Central Nervous Systemt (CNS) stimulants
  Arms: ER stimulant
Other: monitoring — monthly weight, height and BMI checks
  Other Names: monitoring arm
  Arms: weight recovery treatment- monitoring
Other: drug holiday — switch from seven day a week dosing to medication only on school days
  Other Names: Ritalin based product, CNS stimulants
  Arms: weight recovery treatment- drug holiday
Dietary Supplement: caloric supplement — continue current ADHD regimen and add one 8oz liquid caloric supplement at night
  Arms: weight recovery treatment- caloric supplement

SUMMARY:
Previous NIH funded Attention Deficit Hyperactivity Disorder (ADHD) trials in children found that daily stimulant therapy produced sustained growth deficits. However, no federally funded studies have examined the growth suppression associated with modern once a day stimulant medications. Therefore, this study will precisely estimate the risks of stimulant induced growth suppression (SIGS), examine the underlying mechanisms and develop treatments for it. While drug holidays and caloric supplementation are two common treatments for SIGS, there has been little systematic investigation of either. It is unknown if they are effective or feasible. Therefore, using a randomized adaptive design, we will evaluate the efficacy and feasibility of these two practices vs. routine monitoring of growth in 180 prepubertal children with ADHD. An additional 50 subjects will be treated solely with behavioral therapies to evaluate for growth abnormalities associated with ADHD. The study will assess will the risk of SIGS with ER stimulants and the underlying mechanisms while providing evidenced-based treatments for its management.

DETAILED DESCRIPTION:
The study will consist of 4 parts:

1. Screening assessment to determine if a child has ADHD and would be a good candidate to have their ADHD treated with an extended release (ER) stimulant medication. If the answer to step one is yes, then the child will be randomly assigned to receive either medication treatment with an extended release MPH product (OROS MPH). 78% of children with start with this option with 22% assigned to behavioral therapy/counseling treatments for ADHD. There will be no placebo treatments used in this study. All children must be between the ages of 5 and 12 and never have taken stimulant medications for ADHD for more than one week to be eligible for the study.
2. Initial Treatment Phase: The dose of the assigned treatment option will be gradually adjusted over the course of the first 3 months until the child's ADHD is well controlled. If the child is assigned to medication, he/she will start with a low dose of the ER MPH product, and it will be gradually increased until his/her ADHD is in good control. Children assigned to medication will be asked to take it every day of the week for at least the first 6 months. Children assigned to behavior therapy will be asked to avoid using medication for the first 6 months of the study. After month 6 if the first treatment is not effective, the child will be given the chance to try the other option. If any treatment is causing a concerning side effect, he/she can stop taking it at any time and we will provide him/her with other treatment options as part of the study.
3. Ongoing Treatment Phase: We will continue to provide these ADHD treatments for a total of 30 months (2 1/2 years). The dose or type of therapy may be adjusted if needed. The child will be monitored every 1-3 months over this time span. Monitoring includes doctor visits to assess growth and side effects of medication, regular contact with his/her teacher to assess function at school and with you to assess function at home. In total, the child will receive study treatments for approximately 30 months and will be required to come to our center for a minimum of 18 follow up visits over this time. The average visit should take 30 minutes or less.
4. Weight Recovery Phase: Any child whose body mass index or BMI declines by a concerning amount will be randomly assigned to receive 1 of 3 weight promotion treatments to stabilize his/her BMI in order to see if this prevents suppression of height (keeps them growing to be as tall as they should be). We do not expect children assigned to the behavior therapy arm to need these treatments, but the identical weight promotion treatments will be available for children in this group if the need arises.

A) Extra monitoring: A doctor will check the child's growth every month (instead of every 3 months) until his/her BMI has returned to normal.The child will stay on the current daily dose of medication or behavior therapy.

B) Caloric supplementation: Parents will be provided with a flavored calorie drink to give to your child every night and continue on the same daily dose and frequency of medication or behavior therapy. The child will have their growth monitored monthly by a study doctor.

C) Drug Holiday: Participants will now only take medication on school days. Children assigned to behavior therapy will not participate in this treatment as they are not taking any study medication. The child will have their growth monitored monthly by a study doctor.

Once the child's weight recovers, these extra treatments will end and he/she will return to the prior medication treatment (medication7 days a week or behavior therapy) in step 3 and to every 3 month growth assessments. Any time the child's BMI declines again, the extra treatments will restart again.

ELIGIBILITY:
Inclusion Criteria:

* children meeting criteria for any subtype of ADHD between the ages of 5-12 who are stimulant naive

Exclusion Criteria:

* Children who meet any of the following criteria will not be eligible to participate in this study:

  * children with a Full Scale Intelligence Quotient (I below 70 as children with IQs less than this would likely not benefit from the behavior therapy intervention
  * not in full time school or less than 5 or older than 12 years at the time of the screening visit
  * children who have a history of seizures or other neurological problems and are taking medication to prevent seizures as stimulants could worsen seizures
  * children with a history of other medical problems for whom psychostimulant treatment may involve considerable risk including cardiac arrhythmias, hypertension, Tourette's Disorder or history of severe tic exacerbations secondary to stimulant exposure
  * children with a history of other medical problems that could impact appetite or weight such as hypothyroidism, diabetes mellitus, liver or renal disease. Also, children using prescription medication that can significantly impact appetite or weight are excluded
  * children with a childhood history or diagnosis of any of the following mental health disorders: pervasive developmental disorder, schizophrenia or other psychotic disorders, bipolar disorder, post traumatic stress disorder, major depression with serious suicidal thoughts or an eating disorder as stimulants are not safe and effective treatments for these conditions, and these diseases could affect eating habits
  * children whose Body Mass Index is very low (too light for safe use of stimulant medication) or is too high (overweight so not suitable for weight promotion treatments)
  * children allergic to milk proteins as they are in the caloric supplement (lactose intolerance okay)
  * children previously treated with stimulant medications for more than 30 days as this study is focusing on children who have never used stimulant medication before.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2010-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James G Waxmonsky, MD, Principal Investigator — Florida International University
Locations (1):
- Center for Children and Families, Florida International University, Miami, Florida, United States

REFERENCES:
- [Derived] Waxmonsky JG, Pelham WE 3rd, Baweja R, Hale D, Pelham WE Jr. Predictors of Changes in Height, Weight, and Body Mass Index After Initiation of Central Nervous System Stimulants in Children with Attention Deficit Hyperactivity Disorder. J Pediatr. 2022 Feb;241:115-125.e2. doi: 10.1016/j.jpeds.2021.09.030. Epub 2021 Sep 25. PMID 34571023
- [Derived] Baweja R, Waschbusch DA, Pelham WE 3rd, Pelham WE Jr, Waxmonsky JG. The Impact of Persistent Irritability on the Medication Treatment of Paediatric Attention Deficit Hyperactivity Disorder. Front Psychiatry. 2021 Jul 21;12:699687. doi: 10.3389/fpsyt.2021.699687. eCollection 2021. PMID 34366928
- [Derived] Waxmonsky JG, Pelham WE 3rd, Campa A, Waschbusch DA, Li T, Marshall R, Babocsai L, Humphery H, Gnagy E, Swanson J, Hanc T, Fallahazad N, Pelham WE Jr. A Randomized Controlled Trial of Interventions for Growth Suppression in Children With Attention-Deficit/Hyperactivity Disorder Treated With Central Nervous System Stimulants. J Am Acad Child Adolesc Psychiatry. 2020 Dec;59(12):1330-1341. doi: 10.1016/j.jaac.2019.08.472. Epub 2019 Aug 29. PMID 31473291

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavior Therapy: 10 week basic parent training, advanced 8 week parent training course. monthly boosters, option for individual parent training sessions, school consultant assigned to each subject
  behavioral therapy: combination of individual and group parent training plus school consultation
- ER Stimulant: daily use of 12 hour extended release (ER) methylphenidate product
  12 hour methylphenidate product: medication to be taken daily for duration of study unless assigned to weight promotion arm
- Caloric Supplementation: Subjects in either the behavior therapy arm or the medication arm who met criteria for weight recovery were randomly assigned to 1 of 3 weight recovery treatments. This arm consisted of monthly weight checks, continuation of a daily extended release stimulant and the addition of a liquid 8oz caloric supplement every evening.
- Drug Holiday: Subjects in either the behavior therapy arm or the medication arm who met criteria for weight recovery were randomly assigned to 1 of 3 weight recovery treatments. This arm consisted of monthly weight checks and limiting CNS stimulant medication to school days only.
- Monitoring: Subjects in either the behavior therapy arm or the medication arm who met criteria for weight recovery were randomly assigned to 1 of 3 weight recovery treatments. This arm consisted of monthly weight checks and continuation of daily extended release stimulant.
Period: Initial Randomization: ADHD Treatment
Arm/Group | Behavior Therapy | ER Stimulant | Caloric Supplementation | Drug Holiday | Monitoring
Started | 50 | 180 | 0 | 0 | 0
Completed | 32 | 131 | 0 | 0 | 0
Not Completed | 18 | 49 | 0 | 0 | 0
Not completed — Lost to Follow-up | 9 | 35 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 7 | 0 | 0 | 0
Not completed — move away | 2 | 7 | 0 | 0 | 0
Period: Adaptive Randomization: Weight Recovery
Arm/Group | Behavior Therapy | ER Stimulant | Caloric Supplementation | Drug Holiday | Monitoring
Started | 0 | 0 | 24 | 23 | 25
Completed | 0 | 0 | 23 | 20 | 24
Not Completed | 0 | 0 | 1 | 3 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 1
Not completed — moved away | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: all participants assigned to treatment Note that initial randomization was to med or behavior. Those meeting criteria were then adaptively rerandomized to 1 of 3 weight recovery arms.
Groups:
- ER Stimulant: daily use of 12 hour extended release methylphenidate product
  12 hour methylphenidate product: medication to be taken daily for duration of study unless assigned to weight promotion arm
- Total: Total of all reporting groups
Arm/Group | Behavior Therapy | ER Stimulant | Total
Number analyzed (Participants) | 50 | 180 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.54 (2.28) | 8.15 (1.86) | 8.23 (1.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 47 | 61
  Male | 36 | 133 | 169
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 134 | 169
  Not Hispanic or Latino | 15 | 46 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 17 | 22
  White | 45 | 157 | 202
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 180 | 230
zHeight [Mean (Standard Deviation); unit: Z score] | 0.01 (1.00) | 0.09 (0.99) | 0.07 (0.99)
zWeight [Mean (Standard Deviation); unit: Z score] | .350 (.918) | .277 (.912) | 0.314 (0.90)
zBMI [Mean (Standard Deviation); unit: Z score] | 0.581 (0.825) | 0.384 (0.837) | 0.424 (0.85)

OUTCOME MEASURES:

1. Primary Outcome: Change Score for Z-height Baseline to Endpoint
Description: The primary endpoint will be change in z-height at month 30 which is study endpoint.
  Measured as a zscore with more negative units reflecting smaller incremental height gain. Z units used to account for differences between groups in gender and age with both impact height at a fixed time.
Time Frame: month 30 or last assessment point
Population: includes all with 2+ growth assessments from the behavior therapy and ER stimulant arms. Doesn't include adaptive randomization arms (drug holiday, cal supplement, monitoring) as they didn't exist until 2nd randomization. See outcome #10 for change in zht from beginning to end of second randomization.
Measure: Mean (Standard Deviation); unit: Z score
Groups:
- Behavior Therapy: 10 week basic parent training, advanced 8 week parent training course. monthly boosters, option for individual parent training sessions, school consultant assigned to each subject
  behavioral therapy: combination of individual and group parent training plus school consultation
  medication usage allowed after month 6 if still moderately impaired or worse on Clinical Global Impressions
Arm/Group | Behavior Therapy | ER Stimulant
Number analyzed (Participants) | 42 | 170
Z score | -.04 (.46) | -.11 (.41)

2. Secondary Outcome: Change Score for z Weight
Description: difference between baseline and endpoint (month 30 or last assessment point if did not finish study). Measured as a zscore with more negative units reflecting lesser weight gain. Z units used to account for differences between groups in gender and age with both impact weight at a fixed time.
Time Frame: baseline to month 30 or to last assessment point
Population: includes all with 2+ growth assessments from the behavior therapy and ER stimulant arms. Doesn't include adaptive randomization arms (drug holiday, caloric supplement, monitoring) as they did not exist until 2nd randomization. See outcome #11 for change in zwt from beginning to end of second randomization.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Behavior Therapy | ER Stimulant
Number analyzed (Participants) | 42 | 170
Z score | -.01 (.56) | -.19 (.45)

3. Secondary Outcome: Change in zBody Mass Index (BMI)
Description: BMI will be calculated at endpoint (month 30). Difference between baseline and endpoint (month 30 or last assessment point if did not finish study). Measured as a zscore with more negative units reflecting less BMI gain. Z units used to account for differences between groups in gender and age with both impact BMI at a fixed time.
Time Frame: baseline to month 30 or last assessment point
Population: includes all with 2+ growth assessments from the behavior therapy and ER stimulant arms. Doesn't include adaptive randomization arms (drug holiday, caloric supplement, monitoring) as they did not exist until 2nd randomization. See outcome #12 for change in zBMI from beginning to end of second randomization.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Behavior Therapy | ER Stimulant
Number analyzed (Participants) | 42 | 170
Z score | -.06 (.53) | -.21 (.51)

4. Secondary Outcome: Treatment Adherence for Caloric Supplement
Description: percent of days caloric supplement were taken versus prescribed in caloric supplement arm
Time Frame: from entry to exit of caloric supplement arm
Population: those assigned to caloric supplement group
Measure: Mean (Standard Deviation); unit: percentage of days
Groups:
- Weight Promotion Treatment- Caloric Supplement: Subjects in either the behavior therapy arm or the medication arm will be assigned to one of 3 treatments if subject does not meet projected BMI goals- either increased monitoring of growth, caloric supplement or drug holiday where only use ADHD medication for school
  12 hour methylphenidate product: medication to be taken daily for duration of study unless assigned to weight promotion arm
  increased monitoring of growth: monthly weight, height and BMI checks
  drug holiday: switch from seven day a week dosing to medication only on school days
  caloric supplement: continue current ADHD regimen and add one 8oz liquid caloric supplement at night
Arm/Group | Weight Promotion Treatment- Caloric Supplement
Number analyzed (Participants) | 24
percentage of days | 70 (29.4)

5. Secondary Outcome: ADHD Symptoms- Parent Rated
Description: sum of score on 10 item IOWA Conners with range from 0 to 30 and higher values indicating more symptoms. Collected at end point or last assessment point.
Time Frame: at month 30 or last collected assessment point
Population: those assigned to either Behavior therapy or ER stimulant with at least one post baseline assessment of ADHD symptoms. Second randomization arms (drug holiday, cal supplement, monitoring) not included as only relevant outcomes are ht, wt and BMI. All subjects in these arms are either in behavior therapy or er stimulant arm from 1st randomization.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavior Therapy | ER Stimulant
Number analyzed (Participants) | 46 | 175
units on a scale | 15.6 (6.7) | 15.2 (5.7)

6. Secondary Outcome: Change Score for Zheight Months 0 to 6
Description: in addition to the primary outcome of height at month 30, change in z-height from baseline to study month 6 post is also reported. Subjects who were still moderately impaired after 6 months in their initial treatment arm were allowed to cross over and receive the treatments in the other arm so prior to month 6 no participants randomized to behavior arm were prescribed study medication.
  This outcome includes all participants with 2+ growth assessments from the behavior therapy and ER stimulant arms. Doesn't include adaptive randomization arms (drug holiday, cal supplement, monitoring) as they didn't exist until 2nd randomization which did not occur until after this assessment period was over.
  Height converted to z score to account for differences in age and gender. More negative values reflecting smaller incremental height gain.
  If participant dropped out prior to month 6, then the last assessment point was used.
Time Frame: baseline to month 6
Population: participants with at height measurement at month 6
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Behavior Therapy | ER Stimulant
Number analyzed (Participants) | 42 | 170
Z score | 0.00 (0.19) | -0.035 (0.14)

7. Secondary Outcome: ADHD Symptoms- Teacher Rated
Description: sum of items on 10 item IOWA Conners with range from 0-30 and larger values indicating greater symptoms. Collected at endpoint or last assessment point.
Time Frame: month 30 or last assessment point
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavior Therapy | ER Stimulant
Number analyzed (Participants) | 42 | 167
units on a scale | 14.5 (7.2) | 13.8 (7.7)

8. Secondary Outcome: Medication Adherence
Description: % of study days that study ADHD medication was taken when prescribed to be taken; behavior group could be prescribed medication if moderately impaired still after month 6. Once prescribed, all medication was prescribed to be taken 7 days a week except for in the drug holiday weight recovery arm.
Time Frame: denominator is number of days in study for which study med was prescribed
Population: any participants with at least one dose of med prescribed. The second randomization arms are not included as all participants in those arms are derived from these two groups and this assessment period includes the entire duration of the second randomization. Also, the second randomization addressees weight gain, not ADHD treatment.
Measure: Number; unit: % of days dose taken as prescribed
Arm/Group | Behavior Therapy | ER Stimulant
Number analyzed (Participants) | 34 | 122
% of days dose taken as prescribed | 68.1 | 71.1

9. Secondary Outcome: Number of Behavior Therapy Sessions
Description: Raw number of behavior therapy sessions attended; participants could cross over to other treatment arm if moderately impaired after 6 months in initial randomly assigned arm
Time Frame: months 0 through 30
Population: those with at least one follow up assessment. The second randomization arms are not included as all participants in those arms are derived from these two groups and this assessment period includes the entire duration of the second randomization. Also, the second randomization addressees weight gain, not ADHD treatment.
Measure: Mean (Standard Deviation); unit: sessions attended
Groups:
- ER Stimulant: daily use of 12 hour extended release methylphenidate product
  12 hour methylphenidate product: medication to be taken daily for duration of study unless assigned to weight promotion arm Med group allowed to participate in initial basic parent training course Additional Behavioral therapy services allowed after month 6 if still moderately impaired or worse on Clinical Global Impressions
Arm/Group | Behavior Therapy | ER Stimulant
Number analyzed (Participants) | 50 | 174
sessions attended | 8.1 (10.5) | 8.1 (7.3)

10. Secondary Outcome: Change in Height z Score During Weight Recovery Phase (Second Randomization)
Description: difference in height z score from entry into weight recovery phase to exit from weight recovery phase (exact duration varied by participant). Randomization could not occur before month 6 (equaling a 24 month duration) but could start as late as month 29 (equaling a 1 month duration) of treatment based on the pattern of zBMI change by the individual participant.
  Z scores used to account for differences in age and gender. More negative values reflecting less incremental height gain.
Time Frame: between 1 month and 24 months
Population: all participants prescribed an ER stimulant who were also went through the second randomization to one of three weight recovery interventions. One monitoring participant never prescribed med was excluded.First randomization arms not included as not all of those participants had a second randomization as it was adaptively based on change in zBMI.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Caloric Supplementation | Drug Holiday | Monitoring
Number analyzed (Participants) | 24 | 23 | 23
Z score | -0.185 (0.232) | -0.030 (.247) | -0.168 (0.337)

11. Secondary Outcome: Change in Weight z Score During Weight Recovery Phase (Second Randomization)
Description: difference in weight z score from entry into weight recovery phase to exit from weight recovery phase (exact duration varied by participant). Randomization could not occur before month 6 (equaling a 24 month duration) but could start as late as month 29 (equaling a 1 month duration) of treatment based on the pattern of zBMI change by the individual participant.
  Z scores used to account for differences in age and gender. Larger values reflect a greater incremental weight gain.
Time Frame: 1 to 24 months duration
Population: all participants prescribed an ER stimulant who were also went through the second randomization to one of three weight recovery interventions.First randomization arms not included as not all of those participants had a second randomization as it was adaptively based on change in zBMI.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Caloric Supplementation | Drug Holiday | Monitoring
Number analyzed (Participants) | 24 | 23 | 23
Z score | 0.050 (.289) | 0.262 (0.353) | 0.062 (0.331)

12. Secondary Outcome: Change in Zscore for BMI During Weight Recovery Phase (Second Randomization)
Description: difference in BMI z score from entry into weight recovery phase to exit from weight recovery phase (exact duration varied by participant). Randomization could not occur before month 6 (equaling a 24 month duration) but could start as late as month 29 (equaling a 1 month duration) of treatment based on the pattern of zBMI change by the individual participant.
  Z scores used to account for differences in age and gender. Larger values reflecting a greater incremental BMI gain.
Time Frame: between 1 month and 24 months
Population: all participants prescribed an ER stimulant who were also went through the second randomization to one of three weight recovery interventions. First randomization arms not included as not all of those participants had a second randomization as it was adaptively based on change in zBMI.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Caloric Supplementation | Drug Holiday | Monitoring
Number analyzed (Participants) | 24 | 23 | 23
Z score | 0.243 (0.499) | 0.443 (0.459) | 0.247 (0.379)

13. Post Hoc Outcome: Change in Height z Score by Actual Medication Usage
Description: measures change in height z score from baseline to last assessment with participants grouped based on actual medication usage versus randomly assigned group since participants were allowed to cross treatment arms after 6 months and not all participants assigned to medication used it consistently. The rarely med group (n=44) used med <12.5% of the study duration (with most using not at all). The consistent med group (N=38 used) med for at least 87.5% of their time in the study with most using the entire time. The inconsistent med group (N=111), used medication between 12.5 to 87.5 of the time (mean time on med was 45% of the time in the study) The other 37 participants did not have one year of growth data so were excluded from this analysis. Z scores used to account for differences in age and gender between groups. More negative values reflecting a smaller incremental height gain.
Time Frame: baseline to month 30 or last assessment point
Population: Includes all participants with at least one year of growth data as goal was to assess impact of extended treatment on growth. These same outcomes are reported elsewhere for the first randomization arms of Behavior Therapy and Med as well as the second randomization arms of cal supplement, drug holiday and monitoring (see outcomes 1 and 10).
Measure: Mean (Standard Deviation); unit: Z score
Groups:
- Consistent Medication: participants grouped based on actual medication usage versus randomly assigned group since participants were allowed to cross treatment arms after 6 months and not all participants assigned to medication used it consistently. The rarely med group (n=44, 29.5% female) used med <12.5% of the study duration (with most using not at all). The consistent med group used med for at least 87.5% of their time in the study with most using the entire time.
- Inconsistent Medication Group: measures change in z height from baseline to last assessment with participants grouped based on actual medication usage versus randomly assigned group since participants were allowed to cross treatment arms after 6 months and not all participants assigned to medication used it consistently. The inconsistent med group used med at least 12.5% of the time in the study but less than 87.5% of the time in the study (mean usage was 45% of time in study).
- Rare Medication Group: measures change in z height from baseline to last assessment with participants grouped based on actual medication usage versus randomly assigned group since participants were allowed to cross treatment arms after 6 months and not all participants assigned to medication used it consistently. The rare med group used med <12.5% of the study duration (with most using not at all).
Arm/Group | Consistent Medication | Inconsistent Medication Group | Rare Medication Group
Number analyzed (Participants) | 38 | 111 | 44
Z score | -0.248 (.341) | -0.113 (.430) | 0.042 (.464)

14. Post Hoc Outcome: Change in Weight z Score by Actual Medication Usage
Description: measures change in weight z score from baseline to last assessment with participants grouped based on actual medication usage versus randomly assigned group since participants were allowed to cross treatment arms after 6 months and not all participants assigned to medication used it consistently. The rarely med group (n=44) used med <12.5% of the study duration (with most using not at all). The consistent med group (N=38 used med for at least 87.5% of their time in the study with most using the entire time). The inconsistent med group (N=111, 27.5% used medication 45% of the time in the study. The other 37 participants did not have one year of growth data so were excluded from this analysis. Z scores used to account for differences in age and gender between groups. Higher values represent a greater incremental weight gain.
Time Frame: baseline to month 30 or last assessment point
Population: Includes all participants with at least one year of growth data as goal was to assess impact of extended treatment on growth. These same outcomes are reported elsewhere for the first randomization arms of Behavior Therapy and Med as well as the second randomization arms of cal supplement, drug holiday and monitoring (see outcomes 2 and 11).
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Consistent Medication | Inconsistent Medication Group | Rare Medication Group
Number analyzed (Participants) | 38 | 111 | 44
Z score | -0.507 (.335) | -0.177 (.443) | 0.112 (.518)

15. Post Hoc Outcome: Change in BMI z Score by Actual Medication Usage
Description: measures change in BMI z score from baseline to last assessment with participants grouped based on actual medication usage versus randomly assigned group since participants were allowed to cross treatment arms after 6 months and not all participants assigned to medication used it consistently. The rarely med group (n=44) used med <12.5% of the study duration (with most using not at all). The consistent med group (N=38 used med for at least 87.5% of their time in the study with most using the entire time). The inconsistent med group (N=111, 27.5% used medication 45% of the time in the study. The other 37 participants did not have one year of growth data so were excluded from this analysis. Z scores used to account for differences in age and gender between groups. Higher values represent a larger BMI
Time Frame: baseline to month 30 or last assessment point
Population: Includes all participants with at least one year of growth data as goal was to assess impact of extended treatment on growth. These same outcomes are reported elsewhere for the first randomization arms of Behavior Therapy and Med as well as the second randomization arms of cal supplement, drug holiday and monitoring (see outcomes 3 and 12).
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Consistent Medication | Inconsistent Medication Group | Rare Medication Group
Number analyzed (Participants) | 38 | 111 | 44
Z score | -0.554 (.412) | -0.170 (.486) | 0.036 (.528)

16. Post Hoc Outcome: Difference in Height z Score During Weight Recovery Phase (Second Randomization) by Actual Usage
Description: difference in height z score from entry into weight recovery phase to exit from that phase (exact duration varied by participant). Randomization could not occur before month 6 (so max of 24 month duration) but could start as late as month 29 (equaling a 1 month duration) based on the pattern of zBMI change. In this post hoc analysis we grouped participants by what they did (caloric supplementation, drug holiday or monitoring) not what they were randomly assigned to. The most common change was from drug holiday to monitoring for participants who were not using medication on weekends before assignment to drug holiday (family stopped weekend med by own accord prior to 2nd randomization) so assignment to drug holiday did not alter actual frequency of use as was designed to.Therefore they were reclassified as monitoring as frequency of med use did not change.
  Z score used to account for differences in age and gender between groups. Larger values reflect greater height change.
Time Frame: between 1 month and 24 months
Population: all participants using an ER stimulant and were also assigned to a weight recovery arm. Arms from first randomization are not included as not all of those participants progressed to the second randomization which was done adaptively based on change in zBMI. Those arms are reported on for outcome 13.
Measure: Mean (Standard Deviation); unit: Z score
Groups:
- Caloric Supplementation: Subjects in either the behavior therapy arm or the medication arm who met criteria for weight recovery and used caloric supplementation for at least the majority of the days in the weight recovery phase.
  This arm also consisted of monthly weight checks, continuation of a daily extended release stimulant.
- Drug Holiday: Subjects in either the behavior therapy arm or the medication arm who met criteria for weight recovery and were previously using medication on the majority of non school days but then stopped using medication on the majority of non school days.
  This arm also consisted of monthly weight checks and use of ER stimulant on school days only.
- Monitoring: Subjects in either the behavior therapy arm or the medication arm who met criteria for weight recovery and were randomly assigned to 1 of 3 weight recovery treatments and did not change their frequency of medication use after the weight recovery randomization (either used the majority of non school days pre and post randomization or did not use med the majority of non school days pre and post randomization).
  This arm also consisted of monthly weight checks.
Arm/Group | Caloric Supplementation | Drug Holiday | Monitoring
Number analyzed (Participants) | 23 | 16 | 31
Z score | -0.184 (0.238) | -0.095 (0.277) | -0.105 (0.311)

17. Post Hoc Outcome: Change in Weight z Score During Weight Recovery Phase (Second Randomization) Based on Actual Usage
Description: difference in height z score from entry into weight recovery phase to exit from that phase (exact duration varied by participant). Randomization could not occur before month 6 (so max of 24 month duration) but could start as late as month 29 (equaling a 1 month duration) based on the pattern of zBMI change. In this post hoc analysis we grouped participants by what they did (caloric supplementation, drug holiday or monitoring) not what they were randomly assigned to. The most common change was from drug holiday to monitoring for participants who were not using medication on weekends before assignment to drug holiday (family stopped weekend med by own accord prior to 2nd randomization) so assignment to drug holiday did not alter actual frequency of use as was designed to.Therefore they were reclassified as monitoring as frequency of med use did not change.
  Z score used to account for differences in age and gender between groups. Higher values reflect greater incremental weight gain.
Time Frame: between 1 month and 24 months
Population: participants using an ER stimualnt and also randomized to one of the weight recovery treatments. Arms from first randomization are not included as not all of those participants progressed to the second randomization which was done adaptively based on change in zBMI. Those arms are reported on for outcome 14.
Measure: Mean (Standard Deviation); unit: zscore
Arm/Group | Caloric Supplementation | Drug Holiday | Monitoring
Number analyzed (Participants) | 23 | 16 | 31
zscore | 0.055 (0.295) | 0.299 (0.452) | 0.084 (0.265)

18. Post Hoc Outcome: Change in BMI z Score During Weight Recovery Period (Second Randomization) Based on Actual Usage
Description: difference in height z score from entry into weight recovery phase to exit from that phase (exact duration varied by participant). Randomization could not occur before month 6 (so max of 24 month duration) but could start as late as month 29 (equaling a 1 month duration) based on the pattern of zBMI change. In this post hoc analysis we grouped participants by what they did (caloric supplementation, drug holiday or monitoring) not what they were randomly assigned to. The most common change was from drug holiday to monitoring for participants who were not using medication on weekends before assignment to drug holiday (family stopped weekend med by own accord prior to 2nd randomization) so assignment to drug holiday did not alter actual frequency of use as was designed to.Therefore they were reclassified as monitoring as frequency of med use did not change.
  Z score used to account for differences in age and gender between groups. Higher values reflect greater incremental BMI increase.
Time Frame: between 1 month and 24 months
Population: all participants prescribed an ER stimulant and also assigned to one of the weight recovery treatments. Arms from first randomization are not included as not all of those participants progressed to the second randomization which was done adaptively based on change in zBMI. Those arms are reported on for outcome 15.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Caloric Supplementation | Drug Holiday | Monitoring
Number analyzed (Participants) | 23 | 16 | 31
Z score | 0.248 (0.508) | 0.496 (0.576) | 0.260 (.302)

ADVERSE EVENTS:
Time Frame: up to 30 months (max study duration). Population is all participants with at least a baseline side effect rating and at least one additional rating of adverse events post baseline which is 212 cases total. This differs from other enrollment numbers as not all participants assigned to each group completed side effect assessments. We did not want to include missing cases as negative cases (no side effects) as that would impact side effect rates.
Groups:
- Behavior Therapy: Participants completing a baseline assessment and at least one post baseline assessment of adverse events and were initially assigned to behavior arm which included a basic parenting intervention, additional advanced 8 week parent training intervention, monthly boosters, option for individual parent training sessions, and a school consultant assigned to each subject.
  Medication usage allowed after month 6 if at least moderately impaired
  includes all participants with at least one post baseline assessment of adverse events
- ER Stimulant: Participants completing a baseline assessment and at least one post baseline assessment of adverse events who were initially assigned to daily use of extended release CNS Stimulant
  All study medication was prescribed to be taken daily for duration of study unless assigned to weight promotion drug holiday arm
  includes all participants with at least one post baseline assessment of adverse events
- Dose Optimzed: This arm includes the 142 participants that had their dose of study medication systematically optimized through assessment of efficacy and tolerability at home and school. There participants could have come from either of the other two arms- initially assigned to either med or behavior. We added this post hoc arm as a subset of participants randomized to med never used med and a subset of behavior randomized participants did use medication. This group reports adverse event rates only in participants who used med for a sufficient duration to have their dose optimized.
Arm/Group | Behavior Therapy | ER Stimulant | Dose Optimzed
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/171 | 0/136
Serious Adverse Events (participants affected / at risk) | 2/41 | 3/171 | 4/136
Other Adverse Events (participants affected / at risk) | 33/41 | 156/171 | 125/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavior Therapy (N=41) | ER Stimulant (N=171) | Dose Optimzed (N=136)
self injurious behavior (Psychiatric disorders) | 1 (1) | 0 (0) | 1 — child tried to open door in moving car in attempt to harm self. Did lead to psychiatric hospitalization with no further self harm events.
aggression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 — child became defiant towards staff at school and responded with physical aggression when redirected. led to brief psychiatric hospitalization. Event did not recur over course of the study.
appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 — hospitalized for appendectomy
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 — diagnosed with gastroenteritis and hospitalized for one day
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 — diagnosed with pneumonia and hospitalized for treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Behavior Therapy (N=41) | ER Stimulant (N=171) | Dose Optimzed (N=136)
skin picking (Skin and subcutaneous tissue disorders) | 20 | 81 | 57 — measured on Pittsburgh Side Effect Rating Scale
buccal movements (Nervous system disorders) | 10 | 29 | 20 — measured on Pittsburgh Side Effect Rating Scale
anxiety (Psychiatric disorders) | 24 | 104 | 65 — measured on Pittsburgh Side Effect Rating Scale
dull, listless (General disorders) | 10 | 51 | 36 — measured on Pittsburgh Side Effect Rating Scale
headache (Psychiatric disorders) | 12 | 45 | 40 — measured on Pittsburgh Side Effect Rating Scale
stomachache (Gastrointestinal disorders) | 11 | 52 | 43 — measured on Pittsburgh Side Effect Rating Scale
irritability (Psychiatric disorders) | 14 | 80 | 66 — measured on Pittsburgh Side Effect Rating Scale
depressed mood (Psychiatric disorders) | 9 | 55 | 48 — measured on Pittsburgh Side Effect Rating Scale
socially withdrawn (Psychiatric disorders) | 9 | 35 | 27 — measured on Pittsburgh Side Effect Rating Scale
loss of appetite (General disorders) | 16 | 85 | 85 — measured on Pittsburgh Side Effect Rating Scale
trouble sleeping (General disorders) | 11 | 74 | 56 — measured on Pittsburgh Side Effect Rating Scale
motor/verbal tics (Nervous system disorders) | 8 | 30 | 25 — not including buccal movements

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No